CLINICAL TRIAL: NCT04317378
Title: Changes in Temperature in Children Undergoing MRI
Brief Title: Increase in Temperature in Children Undergoing MRI
Acronym: HOT-MR
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Thurid Waagstein Madsen, Nurse anesthetist, Cand scient san student, Rigshospitalet, Denmark
Other Study IDs: TWMADSEN
Record Dates: First submitted 2020-03-09; First posted 2020-03-23 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Magnetic Field Exposure; Temperature Change, Body; Children, Only
Keywords: magnetic resonance Imaging; paediatrics; temperature
MeSH Terms: conditions — Body Temperature Changes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Braun thermoscan /, IRT 6520 — The temperature will be measured in both ears with an ear thermometer. Practically, we will measure the temperature twice when generel anaesthsia is established, and immidiately before and after the MRI scan.

SUMMARY:
An increasing number of children undergo Magnetic Resonance Imaging (MRI). In MRI, radio waves and magnetism are used to form images of the body's interior, to diagnose and monitoring diseases in children. Many children are sedated to be able to collaborate with the MRI procedure. Sedation and general anesthesia cause the child to some extent to lose the ability to regulate his or her own bodytemperature. MRI rooms are most often cold due to the function of the magnet, leading to a risk of hypothermia in young children. Conversely, the MRI scanner generates radio frequencies that are absorbed by the body and converted to heat, which especially in small children due to their large surface area can potentially result in an increase in bodytemperature. In this study we therefore want to investigate changes in bodytemperature in children who are undergoing MRI- scanning within the Neuroanesthesiology Clinic. Furthermore, we want to define possible risk factors for possible temperature changes. Our hypothesis: Children undergoing MRI scanning increase in bodytemperature.

DETAILED DESCRIPTION:
Ear temperature is measured as we are primarily interested in describing temperature changes in the individual child and because this method is less invasive than the alternatives.

ELIGIBILITY:
Inclusion Criteria:

* Age from 12 weeks to 12 years
* Children undergoing MRI scans with the help of anesthesia staff from the Neuroanesthesiology Clinic under general anesthesia or awake
* The children are recruited via prescriptions or the anesthetist immediately before scanning and outside the MRI room. All children who meet the criteria for MRI scan can be included. Acute MRI children, children admitted to intensive care and children who came is directly from the operation if consent is obtained.

Exclusion Criteria:

* Inability at present. and relatives to speak and understand Danish or English. An authorized interpreter may be used for a family that does not have a Danish background and only if written and oral information material is understood otherwise the patient is excluded
* No consent to the study
* Anatomically not possible to measure ear temperature
* Temperature above 39 ° C

Ages: 12 Weeks to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children 12 weeks to 12 years of age undergoing MRI procedure with the assistance of anesthesiologists from the Neuroanesthesiology Clinic may be included. Oral and written consent from the parent or relatives of the child will be obtained in accordance with science ethical rules.
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2020-06-14 (Actual); Study Completion 2020-08-28 (Actual)

PRIMARY OUTCOMES:
Delta temperature ∆Tp = post-temperature - pre-temperature. Delta temperature is defined as the average temperature difference between pre-scan and post scan temperature measurement in right and left ear canal of the child before and after MRI scan. | Ear temperature scan within 5 minuts before and after MRI right outside the MRI suite.
  The average of the temperature measured in the two ear canals is used if the difference is less than 0.5 degrees. If the temperature difference between the two ear canals exceeds 0.5 degrees, it is assumed that the lowest temperature is an error measurement e.g. due to physical block of the ear canal. In that case, the highest temperature measured in one of the two ear canals is used.

SECONDARY OUTCOMES:
Childrens body surface area and temperature increase during MRI | 20 minutes - 3 hours
  Influence on body surface area calculated by weight in kilograms, height in centimeters. For calculation the Du Bois formula is used.
Confounders influence on intervention and temperature outcome | 20 minutes
  Age ( years), height (centimeters ) BMI (kg/m^2) < 18.5 underweight, 18.5 -25 normal weight, > 25 overweight.
MRI | 20 minutes to 3 hours
  Influence of MRI protocol: cerebrum, neuro axis, abdominal, heart and others. MRI duration (minutes) and MRI type (Tesla 1,5 or 3,0)
Influence on body temperature | 5 minutes
  Underlying diseases, infection, fever and use contrast.
  , use of contrast.
Medication | 5 minutes
  Use of paracetamol (acetaminophen) same day of MRI-scanning
External use of cover during MRI | 20 minutes - 3 hours
  Use of blankets to prevent heat loss in babies and children undergoing MRI-scan.

OTHER OUTCOMES:
Anesthesia type and influence on body temperature | 20 minutes - 3 hours.
  Generel anesthesia using propofol infusion or sevoflurane. Sedation or awake during MRI. ASA group 1-4

CONTACTS AND LOCATIONS:
Overall Officials: Thurid W Madsen, RN, Study Director — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Blegdamsvej 9, Copenhagen, Denmark